CLINICAL TRIAL: NCT03816553
Title: SHR-1210, a Novel Anti-pd-1 Antibody, in Combination With Apatinib in Patients With Metastatic, Persistent, or Recurrent Cervical Cancer: a Single-arm, Open Label, Multi-center, Phase II Study
Brief Title: SHR-1210 in Combination With Apatinib in Patients With Metastatic, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-169-01
Record Dates: First submitted 2019-01-13; First posted 2019-01-25 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Recurrent Cervical Carcinoma; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + Apatinib (Experimental): Participants receive SHR-1210 200mg (3mg/kg for underweight patients) intravenously every 2 weeks and apatinib 250mg orally once daily until disease progression or unacceptable toxicity
  Interventions: Drug: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 will be administered as a 30-minute IV infusion Q2W at a dose of 200mg (3mg/kg for underweight patients).
  Other Names: Camrelizumab
Drug: Apatinib — Apatinib will be administered 250mg orally, once daily until progression.
  Other Names: Apatinib Mesylate

SUMMARY:
The purpose of this study is to explore the efficacy and safety of SHR-1210 in combination with apatinib in treating patients with metastatic, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1). Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) selectively inhibits Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2). Patients with metastatic, persistent, or recurrent cervical cancer who failed to first-line chemotherapy +/- bevacizumab will received SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks and apatinib 250mg orally once daily. The efficacy and safety will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy;
2. Age ≥ 18 years and ≤ 70 years;
3. Patients must have measurable disease per RECIST 1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥ 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI),; a lymph node must be ≥ 15 mm in short axis. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy exceeds 3 months;
6. Patients must have had at least one prior systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic carcinoma of the cervix.

   Note: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic carcinoma of the cervix; adjuvant therapy includes cisplatin given concurrent with primary radiation therapy (CCRT) and adjuvant chemotherapy given following the completion of concurrent chemotherapy and radiation therapy
7. Patients must have adequate organ function

   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L
   * Platelet count ≥ 80 × 10^9/L
   * Hemoglobin ≥ 90 g/L
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled)
   * Creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula)
   * Baseline albumin ≥ 28 g/L
   * Thyroid-stimulating hormone (TSH) levels ≤ 1 × ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤ 1 × ULN may be enrolled)
8. Written informed consent.

Exclusion Criteria:

1. Histopathologic diagnoses of tumors other than squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma.
2. Participated in other clinical trials, or finish other clinical trials within 4 weeks.
3. Prior exposure to immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies, or prior exposure to apatinib.
4. Known history of hypersensitivity to any components of the SHR-1210 formulation, or other monoclonal antibody.
5. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
6. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
7. Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association (NYHA) class > 2), unstable or severe angina, severe acute myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.
8. Arterial thrombus or phlebothrombosis within 6 months.
9. Hypertension that can not be well controlled through antihypertensive drugs (systolic pressure ≥ 140 mm Hg and/or diastolic pressure ≥ 90 mm Hg)
10. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
11. Coagulation abnormalities (INR>2.0、PT>16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
12. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events (except for alopecia) due to a previously administered agent.
13. Has known active central nervous system metastases.
14. Patients with a prior invasive malignancy who have had any evidence of disease within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
15. Has an active infection requiring systemic therapy.
16. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
17. Hepatitis B virus (HBV) >2000 IU/ml or DNA ≥ 1×10^4/ml; or hepatitis C virus (HCV) RNA ≥ 1×10^3/ml).
18. Has received a live vaccine within 4 weeks prior to the first dose of trial treatment. Note: Injection of inactivated viral vaccines against seasonal influenza are allowed.
19. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 24 months
  Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression of disease or death from any cause
Overall survival (OS) | Up to approximately 24 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.
6-month PFS rate | From date of enrollment up to 6 months
  The rate of 6-month PFS
9-month OS rate | From date of enrollment up to 9 months
  The rate of 9-month OS
Duration of Response (DCR) | Up to approximately 24 months
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | Up to approximately 24 months
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Incidence of Adverse Events (AEs) in the treatment of SHR1210 in combination with apatinib | Up to approximately 24 months
  Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03.

OTHER OUTCOMES:
Impact of the treatment on Quality of Life (QOL) measured by the Functional Assessment of Cancer Therapy (FACT)-Cervical Trial Outcome of Index (FACT-Cx TOI) | Baseline, every other cycle (each cycle is 28 days) and up to approximately 24 months
  The FACT-Cx TOI is a scale for assessing general QOL of cervical cancer patients consisting of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Cervical Cancer subscale (15 items). Each item in the FACT-Cx TOI was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative statements (or questions), reversal was performed prior to score calculation. The score ranges 0-116 with a large score suggesting better QOL.
Pain assessed by Brief Pain Inventory (BPI) | Baseline, every other cycle (each cycle is 28 days) and up to approximately 24 months
  Single item from the BPI assessing "worst pain" in the past 24 hours, on a 0-10 scale with a higher score indicating more pain than a low score.
PD-L1 expression on tumor and immune cells | Up to approximately 24 months
  The efficacy of the combination of SHR-1210 and apatinib as measured by objective response, will be described in patients according to PD-L1 positive and PD-L1 negative.
Tumor Mutation Burden (TMB) | Up to approximately 24 months
  The impact of TMB on efficacy of the combination of SHR-1210 and apatinib will be explored.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - The First affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Lai Y, Peng H, Yan S, Liu Z, Tong C, Huang X. Multiparametric immune profiling of advanced cervical cancer to predict response to programmed death-1 inhibitor combination therapy: an exploratory study of the CLAP trial. Clin Transl Oncol. 2023 Jan;25(1):256-268. doi: 10.1007/s12094-022-02945-1. Epub 2022 Sep 17. PMID 36115931
- [Derived] Huang X, He M, Peng H, Tong C, Liu Z, Zhang X, Shao Y, Zhu D, Zhang J, Yin JC, Yang F, Lan C. Genomic profiling of advanced cervical cancer to predict response to programmed death-1 inhibitor combination therapy: a secondary analysis of the CLAP trial. J Immunother Cancer. 2021 May;9(5):e002223. doi: 10.1136/jitc-2020-002223. PMID 34011535
- [Derived] Lan C, Shen J, Wang Y, Li J, Liu Z, He M, Cao X, Ling J, Huang J, Zheng M, Zou G, Yan H, Liu Q, Yang F, Wei W, Deng Y, Xiong Y, Huang X. Camrelizumab Plus Apatinib in Patients With Advanced Cervical Cancer (CLAP): A Multicenter, Open-Label, Single-Arm, Phase II Trial. J Clin Oncol. 2020 Dec 1;38(34):4095-4106. doi: 10.1200/JCO.20.01920. Epub 2020 Oct 14. PMID 33052760